CLINICAL TRIAL: NCT02608359
Title: A Prospective, Multicenter, Post-marketing Surveillance to Assess Safety of Zytiga (Abiraterone Acetate Tablets 250 mg) in Indian Patients With Metastatic, Castration Resistant Prostate Cancer as Per Locally Approved Prescribing Information
Brief Title: A Post-marketing Surveillance to Assess Safety of Abiraterone Acetate (Zytiga) in Indian Participants With Metastatic, Castration Resistant Prostate Cancer
Status: Withdrawn | Type: Observational
Why Stopped: No subjects recruited in the study
Sponsor: Johnson & Johnson Private Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: CR107096; 212082PCR4021 (Other: Johnson & Johnson Private Limited)
Record Dates: First submitted 2015-11-17; First posted 2015-11-18 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
Keywords: Post-Marketing Surveillance; Abiraterone Acetate; Zytiga
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Abiraterone Acetate (Zytiga) Post-marketing Surveillance (PMS): This is an observational study and participants will not receive any intervention as a part of this study. All prospective participants who will be prescribed abiraterone acetate tablets 250 milligram (mg) treatment based on independent clinical judgment and as per locally approved prescribing information will be enrolled in the PMS. Participants will be exclusively observed for safety.
  Interventions: Drug: Abiraterone Acetate

INTERVENTIONS:
Drug: Abiraterone Acetate — This is an observational study and participants will not receive any intervention as a part of this study. All prospective participants who will be prescribed abiraterone acetate tablets 250 milligram (mg) treatment based on independent clinical judgment and as per locally approved prescribing information will be enrolled in the PMS. Participants will be exclusively observed for safety.

SUMMARY:
The purpose of this study is to evaluate the safety of abiraterone acetate in Indian participants with metastatic, castration-resistant prostate cancer who have been prescribed abiraterone acetate as per locally approved prescribing information.

DETAILED DESCRIPTION:
This is a prospective (the participants are identified and then followed forward in time for the outcome of the study), multicenter (when more than one hospital or medical school team work on a medical research study), post-marketing surveillance ([PMS], surveillance of drugs, devices, appliances, etc., for efficacy or adverse effects, after they have been released for general sale) study. The study will consist of Screening and Enrolment Visit (Day 1) and Follow-up Period (12 months). For each participant, the follow-up visits will be conducted as per routine clinical practice at month 3, 6 and 9. The End-of-Study (EOS) Visit will be conducted after the completion of 12-months abiraterone acetate (Zytiga) and a telephonic follow-up will be conducted 30 days after the EOS Visit. The total duration of the study will be 13 months. Participants receiving abiraterone acetate as per locally approved prescribing information will be enrolled in the PMS. The use of abiraterone acetate will follow dosing and frequency stipulated in the locally approved prescribing information. Participants will be monitored during treatment of abiraterone acetate and up to 30 days post treatment for collection of adverse events. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with established diagnosis of metastatic castration-resistant prostate carcinoma
* Being newly initiated on Zytiga treatment (abiraterone acetate tablets 250 mg) based on independent clinical judgment of treating physicians as per locally approved prescribing information
* Willing to provide written informed consent indicating that they understand the purpose and are willing to participate in the post-marketing surveillance (PMS)

Exclusion Criteria:

* Participants who are not eligible to receive Zytiga as per the locally approved prescribing information
* Participants participating or planning to participate in any interventional drug trial during the course of this PMS

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Indian participants with metastatic, castration-resistant prostate cancer will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
The Number and Type of Adverse Events Reported by the Investigator or the Patient | up to 13 months
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. The severity of adverse events will be graded using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Private Limited Clinical Trial, Study Director — Johnson & Johnson Private Limited
Locations (3):
- India (3):
  - Bangalore
  - Delhi
  - New Delhi